CLINICAL TRIAL: NCT05668897
Title: A Randomized, Double-blind, Placebo-controlled Single-dose and Multiple-dose Ascending Phase Ia Clinical Trials in Healthy Subjects To Evaluate the Safety, Tolerability and Pharmacokinetics of GST-HG171 Tablets
Brief Title: Safety, Tolerability and Pharmacokinetic Characteristics Evaluation on GST-HG171 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Akeylink Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GST-HG171-I-01
Record Dates: First submitted 2022-12-16; First posted 2022-12-30 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Single-dose ascending group (Experimental): SAD study cotains at least 4 cohorts at dosage of 150mg, 300mg, 600mg and 900mg. Each cohort enrolls 6 subjects receive study drug.
  Interventions: Drug: GST-HG171
- SAD placebo comparator group (Placebo Comparator): SAD study cotains at least 4 cohorts at dosage of 150mg, 300mg, 600mg and 900mg. Each cohort enrolls 2 subjects receive placebo.
  Interventions: Drug: placebo of GST-HG171
- Multi-dose ascending group (Experimental): MAD study cotains 1-3 cohorts which were evaluated in SAD study to be tolerated . Each cohort enrolls 6 subjects receive study drug.
  Interventions: Drug: GST-HG171
- MAD placebo comparator group (Placebo Comparator): MAD study cotains 1-3 cohorts which were evaluated in SAD study to be tolerated . Each cohort enrolls 2 subjects receive placebo.
  Interventions: Drug: placebo of GST-HG171
- Food effect study (Experimental): FE study cotains at least 1 cohort which were evaluated in SAD study to be tolerated . Each cohort enrolls 12 subjects receive study drug on fast or fed condition.
  Interventions: Drug: GST-HG171

INTERVENTIONS:
Drug: GST-HG171 — This study includes single-dose ascending and multiple-dose ascending studies. SAD study contains at least 4 dose groups of 150 mg, 300 mg, 600 mg and 900 mg. MAD study contains 1-3 dose groups which were evaluated in SAD study to be tolerated.
  Arms: Food effect study; Multi-dose ascending group; Single-dose ascending group
Drug: placebo of GST-HG171 — This study includes single-dose ascending and multiple-dose ascending studies. SAD study contains at least 4 dose groups of 150 mg, 300 mg, 600 mg and 900 mg. MAD study contains 1-3 dose groups which were evaluated in SAD study to be tolerated.
  Arms: MAD placebo comparator group; SAD placebo comparator group

SUMMARY:
To Evaluate the Safety, Tolerability and Pharmacokinetics on GST-HG171 Tablets in Randomized, Double-blind, Placebo-controlled Single-dose and Multiple-dose ascending Phase Ia Clinical Trials in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial and fully understand the content, process and possible adverse reactions of the trial;
2. Ability to complete research in accordance with test plan requirements;
3. Subjects (including partners) are willing to take effective pregnancy avoidance measures within 6 months after screening to the last study drug administration;
4. Male and female healthy subjects aged 18 to 50 years (including 18 and 50 years old);
5. Male subjects weigh no less than 50 kg, and female subjects weigh no less than 45 kg. Body mass index (BMI) = body weight (kg) / height 2 (m2), body mass index is in the range of 18 ~ 28 kg / m2 (including critical value);
6. Physical examination, normal or abnormal vital signs have no clinical significance.

Exclusion Criteria:

1. Allergies (multiple drugs and food allergies);
2. Those who smoked more than 5 cigarettes per day in the 3 months before the trial;
3. Have a history of drug abuse and / or alcoholism (drink 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
4. Blood donation or massive blood loss (> 400 mL) within three months before screening;
5. Have a history of dysphagia or any gastrointestinal disease that affects drug absorption, including a history of frequent nausea or vomiting caused by any cause;
6. Have any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis, or gastric and duodenal ulcers;
7. Have taken the study drug or participated in the drug clinical trial within three months before taking the study drug;
8. Have Intended to take any drug that changes the activity of drug metabolizing enzyme 28 days before screening or during the study, including strong inhibitors and inducers that affect the metabolizing enzyme;
9. Took any prescription drugs or herbs within 14 days before screening, or took over-the-counter drugs or any vitamin products within 7 days before screening;
10. Vaccinated within 14 days before screening or planned to be vaccinated during the study;
11. Those who have taken special diets (including dragon fruit, mango, grapefruit, etc.) or have vigorous exercise or other factors affecting drug absorption, distribution, metabolism, excretion, etc. within 2 weeks before screening;
12. Those who cannot tolerate high fat (about 50% of the total calories) and high calorie (about 800~1000 calories) standard meals (only applies to subjects participating in the food effect study);
13. Abnormal ECG has clinical significance;
14. Female subjects were breastfeeding or had a positive serum pregnancy result during the screening period or during the study;
15. Clinical laboratory examinations are abnormal and clinically significant, or find the following diseases with clinical significance (including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, Immune, mental or cardiovascular disease) within 6 months before screening;
16. Positive screening for viral hepatitis (including hepatitis B and C), AIDS antigen / antibody, and Treponema pallidum antibody;
17. Acute disease or concomitant medication occurs from the screening stage to before study medication;
18. Ingested chocolate, any caffeinated or xanthine-rich food or drink 24 hours before taking the study drug;
19. People who have a positive urine drug screen or have a history of drug abuse or have used drugs within the past five years;
20. The investigator believes that there are other subjects who are not suitable for participating in this trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | SAD up to Day 5 and MAD up to Day 9
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Area Under Curve (AUC) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
T1/2 | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Cl/F | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Ae(0~120h) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Fe(0~120h) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Zhou J, Chen H, Mao J, Tang Y, Yan W, Zhang T, Li C, Chen S, Li G, Zhang G, Ding Y, Liu L. Phase I study, and dosing regimen selection for a pivotal COVID-19 trial of GST-HG171. Antimicrob Agents Chemother. 2024 Jan 10;68(1):e0111523. doi: 10.1128/aac.01115-23. Epub 2023 Dec 15. PMID 38099673